CLINICAL TRIAL: NCT06436248
Title: Polygenic Risk Scores and Multi-cancer Early Detection for Ovarian Cancer
Acronym: PROMISE
Status: Active, not recruiting | Type: Observational
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Collaborators: Susan G. Komen Breast Cancer Foundation (Other); Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: UPCC 17824; IRB: 855461 (Other: University of Pennsylvania)
Record Dates: First submitted 2024-04-29; First posted 2024-05-31 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Ovarian Cancer; BRCA Mutation
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The overall goal of the Polygenic Risk Scores and Multi-cancer Early Detection for Ovarian Cancer (PROMISE) study is to better understand how women may incorporate both polygenic risk score (PRS) and novel early detection strategies in their decisions regarding cancer screening and risk reducing surgery. This study will conduct qualitative interviews to better understand women's attitudes regarding polygenic risk score (PRS) and early detection assays.

DETAILED DESCRIPTION:
First, the investigators will conduct qualitative interviews to better understand women's attitudes regarding polygenic risk score (PRS) and early detection assays. Participants will include English-speaking adult women with BRCA1 or BRCA2 pathogenic variants (PV) who have not previously undergone risk-reducing salpingo-oophorectomy (RRSO) (n=24). Interviews will be led by a trained member of the study team using a semi-structured interview guide in order to review definitions of test characteristics (e.g., sensitivity, specificity) and discuss participants' understanding and perceived importance of such test characteristics, and the potential impact of polygenic risk score (PRS) and early detection assay results in informing their cancer prevention decisions. Interviews will be audio-recorded utilizing Zoom audio recording and transcribed using 3Play Media transcription service (Health Insurance Portability and Accountability Act/HIPAA compliant). The investigators will lead analysis of the de-identified transcripts through a process of independent and collaborative thematic content analysis, an established method in qualitative research in order to establish key themes related to clarifying participants' willingness and concerns (e.g., discomfort with test characteristics, perceived ambiguity) for adopting these emerging tests.

Findings from these qualitative interviews will also inform development of hypothetical scenarios that will then be evaluated in a subsequent questionnaire administered to 175-200 English-speaking adult women with BRCA1 or BRCA2 Pathogenic Variants who have not previously undergone risk-reducing oophorectomy or risk-reducing mastectomy. The objective of this survey will be to further evaluate women's decision-making responses to hypothetical polygenic risk score (PRS) and early detection assays, and to determine if there are test characteristics and result thresholds that appear meaningful. Details of this questionnaire and its administration will be included in a future amendment to this current protocol.

Results from year 1 will be used to develop patient materials to use in providing individualized polygenic risk score (PRS) and early detection assay results back to patients in years 2-3. Taken together, investigators hope that this project will provide an estimate on the absolute magnitude of risk which would result in risk reducing surgery within a year, and how a negative early detection assay might modulate such action.

ELIGIBILITY:
Inclusion Criteria:

* Female, age 25 or older (given that women under this age are not generally recommended to receive BRCA1/2 genetic testing)
* Completed full sequence or targeted genetic testing with a clinically confirmed BRCA1 or BRCA2 deleterious mutation identified.
* English-fluent; the surveys and interviews were designed and validated in English and are not currently available in other languages. Translation of questionnaires into other languages would require reestablishing the reliability and validity of these measures. Therefore, participants must be able to communicate in English to complete the surveys.

Exclusion Criteria:

* Previous receipt of any prophylactic oophorectomy
* Personal history of ovarian cancer
* Major psychiatric illness or cognitive impairment that in the judgment of the study investigators would preclude study participation.
* Any patients who are unable to comply with the study procedures as determined by the study investigators or study staff.

Min Age: 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Target population is women, age 25 or over, with likely pathogenic or pathogenic variants in BRCA1 or BRCA2 and no personal history of ovarian cancer or risk-reducing oophorectomy surgery.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
To assess how women will use information regarding polygenic risk score (PRS) and early detection assays to inform prophylactic surgery decisions through interviews | 1 year
  The investigators will assess how women will use information regarding polygenic risk score (PRS) and early detection assays to inform prophylactic surgery decisions through semi-structured interviews and thematic content analyses.

CONTACTS AND LOCATIONS:
Overall Officials: Susan Domchek, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- Abramson Cancer Center, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No